CLINICAL TRIAL: NCT04803916
Title: Pre-stenotic Inflammation Following Endoscopic Balloon Dilatation in Crohn's Disease: A Prospective Study
Status: Recruiting | Type: Observational
Sponsor: Shaare Zedek Medical Center (Other)
Collaborators: Sheffield Children's NHS Foundation Trust (Other); Bambino Gesù Hospital (Unknown); University of Roma La Sapienza (Other); Hopital Universitaire Robert-Debre (Other)
Responsible Party: Principal Investigator, Oren Ledder, MD, Principal Investigator, Shaare Zedek Medical Center
Other Study IDs: Inflammation following EBD
Record Dates: First submitted 2020-08-31; First posted 2021-03-18 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Crohn Disease
Keywords: Crohn; Stricture; Endoscopic Balloon Dilatation
MeSH Terms: conditions — Crohn Disease; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As a consequence of chronic relapsing inflammation in Crohn's disease (CD), progressive bowel damage and scarring occurs in affected regions of intestine. This damage often leads to narrowing, or stricturing of the bowel lumen, and even complete bowel obstruction. Stricturing CD is thought to be a major contributor to penetrating complications including abscesses and fistulae.

Depending on the severity and clinical significance of fixed strictures, treatment options include either endoscopic balloon dilatation (EBD), or surgery with either resection or stricturoplasty recommended on a case-by-case basis.

EBD has been shown to be a safe alternative to surgery in management of CD strictures.

While the short- and medium-term clinical outcomes of EBD have been well described, less well studied is the impact of relieving Crohn's strictures on the inflammatory load proximal to the stricture. The restricted flow of fecal contents through a stricture creates a region of relative stasis in the bowel loops immediately proximal to the stricture, appreciated at times by pre-stenotic dilatation on cross-sectional imaging. This stasis fosters localized bacterial overgrowth and worsening dysbiosis in these bowel loops.

The investigators hypothesize that improvement of fecal flow by way of successful balloon dilatation of a CD stricture, could independently reduce the inflammatory burden, not only in the stenotic segment but also in the proximal loop of bowel.

DETAILED DESCRIPTION:
This prospective, observational study will include both pediatric and adult patients with stricturing CD on stable therapy who are planned to undergo EBD for management of a Crohn's stricture.

Included patients are those in whom the treating physician is planning a colonoscopic EBD for a CD stricture. Patients will be followed with imaging, clinical assessment, serologic testing, stool microbiome and endoscopic assessment at time of EBD, and post-EBD. EBD will be performed to a target dilatation size of 18-20mm. If the stricture is deemed too narrow to allow dilatation to target size in a single session, graduated dilatations at a number of sessions can be undertaken at the treating clinician discretion. Time-point of week 0 will be defined as achievement of dilatation target size.

Clinical assessment, blood and stool for calprotectin and microbiome, and focused bowel US to be performed within a 4 week period prior to EBD. Previous imaging (US/MRE/CTE) from 2-4 months prior to EBD, where performed, will also be assessed.

In the absence of any contra-indication, repeat colonoscopy will be performed at week 12 (±2 weeks) to assess stricture size and assess extent of mucosal inflammation at the stricture site and the pre-stenotic region. Follow-up clinical review with repeat blood tests, stool for calprotectin and microbiome and focused bowel US will also be performed at week 12 (±2 weeks).

Endoscopic images from pre-stenotic bowel loop and bowel US from week 0 and week 12 will be centrally read by two central readers blinded to the patient and stage. An average of pre-stenotic region SES-CD score and US-derived outcome measures from both readers will be recorded. Where available, imaging from 2-4 months pre-EBD, either US, MRE or CTE, will be assessed by the same central readers.

Patients in whom successful balloon dilatation was achieved (see definitions below) will be included in the primary analysis. Patients in whom dilatation was attempted but was not successful (see below) will also be followed and will be analyzed as control group.

Patient's medications are to remain unchanged throughout the follow-up period, including biologic type or dose, or addition of corticosteroids/nutritional therapy, unless the treating physician decides otherwise on clinical grounds, in which case the patient will be defaulted from analysis. Patients on corticosteroid or nutritional therapy at recruitment can continue to wean therapy as per clinician directive.

ELIGIBILITY:
Inclusion criteria:

* Patients diagnosed with CD as per most recent international guidelines.
* Presence of strictured bowel (jejunal, ileal, colonic or ileocecal valve), either primary or anastomotic in nature, with prestenotic dilatation >2.5cm loop diameter as demonstrated on cross-sectional imaging (Magentic Resonance Enteroclysis (MRE), Computerized Tomography Enteroclysis (CTE) or ultrasound (US))
* Evidence of pre-stenotic inflammation defined as wall thickness ≥5mm on cross-sectional imaging, or pre-stenotic SES-CD ≥3.
* Planned EBD as per clinical management.
* Unchanged CD medications - 3 months no change in therapy including immunomodulators (thiopurines or methotrexate), biological therapies, corticosteroid therapy, or nutritional therapy with exclusive enteral nutrition (EEN) or partial enteral nutrition (PEN).
* No planned treatment changes or additions over the 3 months following recruitment. The treating physician can change treatment at any time should the clinical need arise however the patient will be excluded from primary analysis

Exclusion criteria:

* Any patient deemed not appropriate for EBD by treating physician due to stricture- specific, or patient-specific reasons will not be included
* Change in therapy (dose or type) in the 3 months prior to planned EBD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This prospective, observational study will include both pediatric and adult patients with stricturing CD on stable therapy who are planned to undergo EBD for management of a Crohn's stricture.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Endoscopic response | 12 weeks compared to week 0
  Decrease in SES-CD in the pre-stenotic region of ≥ 3 at 12 weeks compared to week 0

SECONDARY OUTCOMES:
Endoscopic healing | week 12
  Post-endoscopic balloon dilatation (EBD) mucosal healing in pre-stenotic region defined as regional SES-CD ≤ 1
Wall thickness | week 12 compared to week 0
  ≥30% reduced intestinal wall thickness in pre-stenotic loop of bowel 12 weeks following successful EBD
Limberg score US | week 12 compared to week 0
  Decrease in Limberg grade of hyperemia in pre-stenotic region of ≥ 2
Luminal diameter | week 12 compared to week 0
  >50% reduction of ratio of maximal upstream luminal diameter to minimal downstream luminal diameter
Inflammed length | week 12 compared to week 0
  >50% reduced length of involved pre-stenotic inflamed region
Obstructive score reduction | week 12
  CDOS ≤ 1 at week 12
Clinical remission | week 12
  Clinical remission as measured by physician global assessment (PGA). 0-100 mm scale 0 being full remission (lower score better outcome)
Stool calprotectin | week 12 compared to week 0
  >50% reduction in stool calprotectin at week 12
No treatment escalation | week 12
  No treatment escalation following EBD
Comparison of imaging and calprotectin | week 12
  Comparison of outcome measures from cross-sectional imaging and stool calprotectin at week 12 between patients with successful EBD vs those with unsuccessful EBD "control".
Clinical remission | week 12
  Clinical remission as measured by Crohn's Disease Activity Index (CDAI )< 150 at week 12.Lower score better outcome
Clinical remission | week 12
  Clinical remission as measured by wPCDAI < 12.5 at week 12

CONTACTS AND LOCATIONS:
Overall Officials: Oren Ledder, Principal Investigator — Department of Gastroenterology and Nutrition, Shaare Zedek Medical Center, Jerusalem, Israel
Locations (1):
- Shaare Zedek, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided